CLINICAL TRIAL: NCT03056027
Title: Evaluation of the Impact of Open or Laparoscopic Preperitoneal Inguinal Hernia Repair on Arterial and Venous Testicular Vascularization by Means of Ecocolordoppler Ultrasound Examination
Brief Title: Testicular Vascular Evaluation in Patients Undergoing Inguinal Hernia Repair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, acestari, Head Department of Urology, Istituto Auxologico Italiano
Other Study IDs: IAI - URO/CHIR - TEP/OPEN
Record Dates: First submitted 2017-02-11; First posted 2017-02-16 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Inguinal Hernia; Testicular Diseases
MeSH Terms: conditions — Hernia, Inguinal; Testicular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Open: Patient submitted to open inguinal hernia repair
  Interventions: Diagnostic Test: Ecocolordoppler ultrasound testicular evaluation
- Group extraperitoneal laparoscopic: Patients submitted to total extraperitoneal laparoscopic inguinal hernia repair
  Interventions: Diagnostic Test: Ecocolordoppler ultrasound testicular evaluation

INTERVENTIONS:
Diagnostic Test: Ecocolordoppler ultrasound testicular evaluation — Ecocolordoppler ultrasound testicular evaluation

SUMMARY:
Patients scheduled to undergo laparoscopic preperitoneal or open inguinal hernia repair will be evaluated by means of scrotal/testicular ecocolordoppler ultrasound investigation before and after surgery in order to rule out the potential impact of the surgical procedure on testicular arterial and venous blood flow

DETAILED DESCRIPTION:
Patients scheduled to undergo laparoscopic preperitoneal or open inguinal hernia repair will be evaluated by means of scrotal/testicular ecocolordoppler ultrasound investigation before and after surgery in order to rule out the potential impact of the surgical procedure on testicular arterial and venous blood flow

Ecocolordoppler will evaluate:

1. testicular arterial flow (Peak Systolic Velocity Testicular Artery - End-Diastolic Velocity Testicular Artery - Resistive Index testicular Artery)
2. venous impaired outflow using varicocele classifications (DUBIN - scale 1-3; HIRSCH scale 1-5)
3. testicular volume

ELIGIBILITY:
Inclusion Criteria:

* Inguinal hernia with surgical indication for surgical repair

Exclusion Criteria:

* History of urologic surgery and/or radiotherapy
* Recurrence of inguinal hernia

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by inguinal hernia, scheduled to undergo either open or laparoscopic extraperitoneal inguinal hernia repair
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2017-10-30 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes in arterial and venous testicular vascularization before and after inguinal hernia repair | Preoperatively - 1 and 4 months after surgery
  evaluation testicular of arterial and venous blood flow by means of ecocolordoppler ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cestari, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Andrea Cestari, Milan, Italy

IPD SHARING:
Plan to Share IPD: No